CLINICAL TRIAL: NCT03821545
Title: The Immunomodulatory Effects of Ketamine and Lidocaine in Abdominal Surgery: Double-Blind, Placebo-Controlled Clinical Study
Brief Title: The Anti-inflammatory Effect of Anesthetics in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Helena Ostovic, Helena Ostovic MD, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Ostovic
Record Dates: First submitted 2018-12-28; First posted 2019-01-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: Anti-Inflammatory Effect; Surgical Stress; Lidocaine; Ketamine; Abdominal Surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine Group (Active Comparator)
  Interventions: Other: Lidocaine
- Ketamine Group (Active Comparator)
  Interventions: Other: Ketamine
- Lidocaine and Ketamine Group (Active Comparator)
  Interventions: Other: Lidocaine and Ketamine
- Placebo (0.9% NaCl) Group (Placebo Comparator)
  Interventions: Other: Placebo (0.9% NaCl)

INTERVENTIONS:
Other: Lidocaine — Lidocaine will be administered at a dose of 1.5 mg/kg prior to surgical incision followed by an infusion at a rate of 1.5-2 mg/kg/hr until the end of surgery.
  Arms: Lidocaine Group
Other: Ketamine — Ketamine will be administered at a dose of 0.5 mg/kg in a bolus prior to surgical incision followed by an infusion at a rate of 0.1-0.2 mg/kg/hr until the end of surgery.
  Arms: Ketamine Group
Other: Lidocaine and Ketamine — Lidocaine will be administered at a dose of 1.5 mg/kg prior to surgical incision followed by an infusion at a rate of 1.5-2 mg/kg/hr until the end of surgery. Ketamine will be administered at a dose of 0.5 mg/kg in a bolus prior to surgical incision followed by an infusion at a rate of 0.1-0.2 mg/kg/hr until the end of surgery.
  Arms: Lidocaine and Ketamine Group
Other: Placebo (0.9% NaCl) — Bolus and continuous placebo infusion (0.9% NaCl) will be equally administered at the same dose as the aforementioned anesthetics until the end of the surgery.
  Arms: Placebo (0.9% NaCl) Group

SUMMARY:
Clinical studies have shown that IV administration of anesthetics, lidocaine and ketamine with their anti-inflammatory properties, modulates the acute immune response associated with surgical tissue injury, and in this manner they are able to reduce postoperative pain. Lidocaine has anti-inflammatory effects on polymorphonuclear granulocytes, IL-6 and IL-8 cytokines, complement component C3a and IL-1ra in serum. Ketamine produces its anti-inflammatory effects by reducing CRP and IL-6 in serum and by inhibiting NF-kB, which regulates gene transcription responsible for the production of proinflammatory factors.

Perioperative combinend IV administration of lidocaine and ketamine could have a more favorable anti-inflammatory effect compared to anesthetic given alone or with placebo.

To investigate the effects of lidocaine and ketamine in patients undergoing abdominal surgery on: acute immune response following the level of proinflammatory factors in serum (CRP, IL-6, IL-8); postoperative pain management; recovery of bowel function; administration of opioids; reduction of total treatment costs; length of hospital stay (LOHS)

A double-blind, placebo-controlled study will include 100 patients undergoing open colorectal surgery. Patients will be randomly assigned to one of four groups: lidocaine, ketamine, lidocaine-ketamine, and placebo. Lidocaine will be administered at a dose of 1.5 mg/kg prior to surgical incision followed by an infusion at a rate of 1.5-2 mg/kg/hr until the end of surgery. Ketamine will be administered at a dose of 0.5 mg/kg in a bolus prior to surgical incision followed by an infusion at a rate of 0.1-0.2 mg/kg/hr until the end of surgery. Bolus and continuous placebo infusion (0.9% NaCl) will be equally administered at the same dose as the aforementioned anesthetics until the end of the surgery.

Proinflammatory markers in serum (CRP, IL-6, IL-8) will be measured before induction of anesthesia, then 12 hours and 36 hours following the completion of surgery. The intensity of pain will be measured using the VAS score 2 hours and 4 hours following surgery and every 12 hours the following days. The investigators will measure also the consumption of opioids during and after surgery, the length of stay in the ICU, where pain control and analgesics use will be measured, as well as recovery of bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery
* Expected duration of the operation > 2 hours

Exclusion Criteria:

* Patients ≤ 18 years of age
* Patients with history of allergy to local anesthetics
* Chronic opioid analgesic
* Patients who are unwilling or unable to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Concentration of inflammatory markers | 1-2 days
  Measuring of inflammatory markers in serum (CRP, IL-6, IL-8) before induction of anesthesia, then 12 hours and 36 hours following the completion of surgery

SECONDARY OUTCOMES:
Opioid consumption during anesthesia | 1 day
  Measuring of total opioid consumption during intraoperative period
VAS- scores | 2 days
  Measuring pain scores VAS scores 2 hours and 4 hours following surgery and every 12 hours the following 2 days.
Analgesic consumption | 2 days
  Measuring total analgesic consumption for 48 hours following the completion of surgery
Recovery of bowel function | 1-5 days
  Measuring time to firs bowel movement
Length of hospital stay | 1- 30 days
  Follow-up patients until hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The Anti-inflammatory Effect of Anesthetics in Abdominal Surgery, Zagreb, Croatia

REFERENCES:
- [Derived] Ostovic H, Simac B, Prazetina M, Bradic N, Persec J. The Effect of Intravenous Lidocaine, Ketamine, and Lidocaine-Ketamine Combination in Colorectal Cancer Surgery: A Randomized Controlled Trial. Anesth Analg. 2025 Jan 1;140(1):67-76. doi: 10.1213/ANE.0000000000006555. Epub 2023 May 24. PMID 37224065